CLINICAL TRIAL: NCT04867785
Title: A Phase 2 Study of Once-Weekly LY3437943 Compared With Placebo and Dulaglutide in Participants With Type 2 Diabetes
Brief Title: A Study of LY3437943 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17774; J1I-MC-GZBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — retatrutide; dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 0.5 milligrams (mg) LY3437943 (Experimental): Participants received 0.5 mg LY3437943 administered as SC (subcutaneous) injection once weekly (QW).
  Interventions: Drug: LY3437943
- 4 mg LY3437943 (2 mg) (Experimental): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 4 mg LY3437943 (4 mg) (Experimental): Participants received 4 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 8 mg LY3437943 (2 mg) (Experimental): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943 and then 8 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 8 mg LY3437943 (4 mg) (Experimental): Participants received 4 mg LY3437943 starting dose followed by 8 mg LY3437943 administered as a SC injection QW.
  Interventions: Drug: LY3437943
- 12 mg LY3437943 (2 mg) (Experimental): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943, then 8 mg LY3437943, then 12 mg LY3437943 administered as a SC injection QW.
  Interventions: Drug: LY3437943
- 1.5 mg Dulaglutide (Active Comparator): Participants received 1.5 mg dulaglutide administered as SC single-dose pen injection QW.
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): Participants received placebo administered as SC injection QW.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: 0.5 milligrams (mg) LY3437943; 12 mg LY3437943 (2 mg); 4 mg LY3437943 (2 mg); 4 mg LY3437943 (4 mg); 8 mg LY3437943 (2 mg); 8 mg LY3437943 (4 mg)
Drug: Dulaglutide — Administered SC
  Arms: 1.5 mg Dulaglutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of LY3437943 in participants with type 2 diabetes (T2D) who failed to achieve adequate glycemic control on diet and exercise alone or on a stable dose of metformin. This study will last about 43 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have an HbA1c value at screening of ≥7.0% and ≤10.5% and treated with diet and exercise alone or with a stable dose of metformin (either immediate release or extended release, 1000 milligram (mg)/day and not more than the locally approved dose) for at least 3 months prior to screening.

Exclusion Criteria:

* Have type 1 diabetes mellitus (T1DM)
* Have ketoacidosis
* Have retinopathy, maculopathy
* Have history of pancreatitis
* Have obesity induced by other endocrine disorders
* Have uncontrolled hypertension
* Have acute or chronic hepatitis
* Have chronic kidney disease
* Have an autoimmune abnormality for example, lupus or rheumatoid arthritis
* Have an active or untreated malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (43):
- United States (40):
  - Syed Research Consultants Llc, Sheffield, Alabama
  - San Fernando Valley Health Institute, Canoga Park, California
  - Valley Endocrine, Fresno, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - Catalina Research Institute, LLC, Montclair, California
  - National Research Institute - Panorama City, Panorama City, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - National Research Institute (NRI) - Santa Ana, Santa Ana, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - South Florida Clinical Research Institute, Margate, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Elite Clinical Trials, Blackfoot, Idaho
  - Humphreys Diabetes Center, Boise, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Elite Clinical Trials, Rexburg, Idaho
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Centennial Medical Group, Elkridge, Maryland
  - MediSync Clinical Research, Petal, Mississippi
  - Clinvest Research LLC, Springfield, Missouri
  - Logan Health Research, Kalispell, Montana
  - Lillestol Research, Fargo, North Dakota
  - Intend Research, LLC, Norman, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - The Research Center of The Upstate, Greenville, South Carolina
  - Dallas Diabetes Research Center, Dallas, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Laila A Hassan, MD, PA, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - Universal Research Group, Tacoma, Washington
  - The Vancouver Clinic, Vancouver, Washington
- Puerto Rico (3):
  - Advanced Clinical Research, LLC, Bayamón
  - Manati Center for Clinical Research, Manatí
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Coskun T, Wu Q, Schloot NC, Haupt A, Milicevic Z, Khouli C, Harris C. Effects of retatrutide on body composition in people with type 2 diabetes: a substudy of a phase 2, double-blind, parallel-group, placebo-controlled, randomised trial. Lancet Diabetes Endocrinol. 2025 Aug;13(8):674-684. doi: 10.1016/S2213-8587(25)00092-0. Epub 2025 Jun 30. PMID 40609566
- [Derived] Rosenstock J, Frias J, Jastreboff AM, Du Y, Lou J, Gurbuz S, Thomas MK, Hartman ML, Haupt A, Milicevic Z, Coskun T. Retatrutide, a GIP, GLP-1 and glucagon receptor agonist, for people with type 2 diabetes: a randomised, double-blind, placebo and active-controlled, parallel-group, phase 2 trial conducted in the USA. Lancet. 2023 Aug 12;402(10401):529-544. doi: 10.1016/S0140-6736(23)01053-X. Epub 2023 Jun 26. PMID 37385280
- See also: A Study of LY3437943 in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/6tv02tRhvMamBP866x6OPm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four maintenance doses of LY3437943 were evaluated: 0.5 mg, 4 mg, 8 mg, and 12 mg. Dose escalation occurred in certain cohorts up to Week 12 during the 36-week treatment period. For maintenance doses equal to or greater than 4 mg, the initial dose will be 2 mg or 4 mg followed by additional escalation steps as appropriate.
Groups:
- Placebo: Participants received placebo administered as subcutaneous (SC) injection once weekly (QW).
- 1.5 Milligrams (mg) Dulaglutide: Participants received 1.5 mg dulaglutide administered as SC single-dose pen injection QW.
- 0.5 mg LY3437943: Participants received 0.5 mg LY3437943 administered as SC injection QW.
- 12 mg LY3437943 (2 mg): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943, then 8 mg LY3437943, then 12 mg LY3437943 administered as SC injection QW.
Period: Overall Study
Arm/Group | Placebo | 1.5 Milligrams (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Started | 45 | 46 | 47 | 23 | 24 | 26 | 24 | 46
Received at Least 1 Dose of Study Drug | 45 | 46 | 47 | 23 | 24 | 26 | 24 | 46
Completed | 34 | 40 | 41 | 19 | 21 | 25 | 22 | 35
Not Completed | 11 | 6 | 6 | 4 | 3 | 1 | 2 | 11
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 4 | 4 | 3 | 2 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 2 | 2 | 1 | 2 | 0 | 2 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Inadvertent Enrollment | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Eligibility Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- 8 mg LY3437943 (4 mg): Participants received 4 mg LY3437943 starting dose followed by 8 mg LY3437943 administered as SC injection QW.
- Total: Total of all reporting groups
Arm/Group | Placebo | 1.5 mg Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg) | Total
Number analyzed (Participants) | 45 | 46 | 47 | 23 | 24 | 26 | 24 | 46 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.56 (10.83) | 54.94 (10.45) | 57.21 (9.69) | 57.70 (8.14) | 57.58 (10.00) | 57.00 (7.37) | 53.83 (9.03) | 54.37 (9.72) | 56.19 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 33 | 23 | 8 | 12 | 16 | 15 | 26 | 156
  Male | 22 | 13 | 24 | 15 | 12 | 10 | 9 | 20 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 27 | 9 | 13 | 12 | 9 | 20 | 131
  Not Hispanic or Latino | 23 | 26 | 20 | 14 | 10 | 14 | 15 | 26 | 148
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Asian | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 6 | 1 | 2 | 3 | 4 | 3 | 33
  White | 36 | 36 | 40 | 20 | 22 | 23 | 20 | 38 | 235
  More than one race | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 45 | 46 | 47 | 23 | 24 | 26 | 24 | 46 | 281
Percentage of Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.39 (1.139) | 8.22 (0.919) | 8.35 (1.172) | 8.07 (0.870) | 8.20 (1.207) | 8.34 (1.120) | 8.20 (1.261) | 8.28 (1.066) | 8.27 (1.086)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: Change in HbA1c (%) from baseline in LY3437943 relative to placebo. HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least squares (LS) mean was calculated using mixed model repeated measures (MMRM) for post-baseline measures: Variable = Treatment*Time + Strata*Time + Baseline*Time.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants with baseline and post-baseline value at the specified time point excluding participants discontinuing study drug due to inadvertent enrollment and data after permanent discontinuation of study drug or initiation of rescue medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | 1.5 mg Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
percentage of HbA1c | -0.05 (0.21) | -1.41 (0.12) | -0.43 (0.20) | -1.39 (0.14) | -1.30 (0.22) | -1.99 (0.15) | -1.88 (0.21) | -2.01 (0.11)
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.188, Mixed Models Analysis; Least Squares (LS) Mean Difference = -0.38, 95% CI 2-sided [-0.94 to 0.18]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.34, 95% CI 2-sided [-1.84 to -0.85]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.25, 95% CI 2-sided [-1.85 to -0.65]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.94, 95% CI 2-sided [-2.44 to -1.43]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.83, 95% CI 2-sided [-2.42 to -1.24]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.96, 95% CI 2-sided [-2.43 to -1.50]

2. Secondary Outcome: Change From Baseline in HbA1c
Description: Change in HbA1c (%) from baseline in LY3437943 relative to dulaglutide. LSMean was calculated using MMRM for post-baseline measures: Variable = Treatment*Time + Strata*Time + Baseline*Time.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- 1.5 Milligram (mg) Dulaglutide: Participants received 1.5 mg dulaglutide administered as SC single-dose pen injection QW.
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
percentage of HbA1c | -0.05 (0.21) | -1.41 (0.12) | -0.43 (0.20) | -1.39 (0.14) | -1.30 (0.22) | -1.99 (0.15) | -1.88 (0.21) | -2.01 (0.11)
Statistical Analysis 1: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 0.98, 95% CI 2-sided [0.52 to 1.43]
Statistical Analysis 2: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.935, Mixed Models Analysis; LSMean Difference = 0.01, 95% CI 2-sided [-0.34 to 0.37]
Statistical Analysis 3: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.668, Mixed Models Analysis; LSMean Difference = 0.11, 95% CI 2-sided [-0.39 to 0.60]
Statistical Analysis 4: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p = 0.002, Mixed Models Analysis; LSMean Difference = -0.58, 95% CI 2-sided [-0.95 to -0.21]
Statistical Analysis 5: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.056, Mixed Models Analysis; LSMean Difference = -0.47, 95% CI 2-sided [-0.95 to 0.01]
Statistical Analysis 6: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.61, 95% CI 2-sided [-0.93 to -0.29]

3. Secondary Outcome: Change From Baseline in HbA1c
Description: Change in HbA1c (%) from baseline in LY3437943 relative to placebo and dulaglutide. LSMean was calculated using MMRM for post-baseline measures: Variable = Treatment*Time + Baseline HbA1c Group (<=8.5%, >8.5%)*Time + Baseline Body Mass Index (BMI) Group (<30 kilograms/square meter (kg/m2), >=30 kg/m2)*Time + Baseline*Time.
Time Frame: Baseline, 36 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
percentage of HbA1c | -0.30 (0.24) | -1.36 (0.13) | -0.54 (0.20) | -1.30 (0.20) | -1.50 (0.19) | -2.13 (0.17) | -1.93 (0.22) | -2.16 (0.13)
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.448, Mixed Models Analysis; LSMean Difference = -0.24, 95% CI 2-sided [-0.85 to 0.38]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = -0.99, 95% CI 2-sided [-1.60 to -0.38]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.20, 95% CI 2-sided [-1.80 to -0.59]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.83, 95% CI 2-sided [-2.41 to -1.24]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.63, 95% CI 2-sided [-2.27 to -0.99]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.85, 95% CI 2-sided [-2.39 to -1.31]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 0.82, 95% CI 2-sided [0.35 to 1.29]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.796, Mixed Models Analysis; LSMean Difference = 0.06, 95% CI 2-sided [-0.41 to 0.53]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.548, Mixed Models Analysis; LSMean Difference = -0.14, 95% CI 2-sided [-0.61 to 0.32]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.77, 95% CI 2-sided [-1.19 to -0.36]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.025, Mixed Models Analysis; LSMean Difference = -0.57, 95% CI 2-sided [-1.08 to -0.07]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.80, 95% CI 2-sided [-1.16 to -0.44]

4. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0%
Description: Percentage of participants reaching HbA1c <7.0% in LY3437943 relative to placebo and dulaglutide. Estimated percentage was determined by logistic regression model with an intercept term, treatment group, baseline BMI stratum [<30 kg/m2, ≥30 kg/m2] as fixed effects, and baseline HbA1c value as a covariate.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
percentage of participants | 18 | 52 | 32 | 53 | 66 | 88 | 78 | 86
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.121, Regression, Logistic; Risk Difference (RD) = 0.14, 95% CI 2-sided [-0.04 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.002, Regression, Logistic; Risk Difference (RD) = 0.36, 95% CI 2-sided [0.13 to 0.59]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.48, 95% CI 2-sided [0.28 to 0.68]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.70, 95% CI 2-sided [0.53 to 0.87]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.60, 95% CI 2-sided [0.39 to 0.82]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.68, 95% CI 2-sided [0.51 to 0.85]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p = 0.030, Regression, Logistic; Risk Difference (RD) = -0.21, 95% CI 2-sided [-0.39 to -0.02]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.938, Regression, Logistic; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.22 to 0.24]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.209, Regression, Logistic; Risk Difference (RD) = 0.13, 95% CI 2-sided [-0.07 to 0.33]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.35, 95% CI 2-sided [0.18 to 0.53]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.024, Regression, Logistic; Risk Difference (RD) = 0.26, 95% CI 2-sided [0.03 to 0.48]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.33, 95% CI 2-sided [0.16 to 0.51]

5. Secondary Outcome: Percentage of Participant Reaching HbA1c <7.0%
Description: as for outcome 4
Time Frame: Week 36
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
percentage of participants | 22 | 60 | 37 | 61 | 59 | 82 | 78 | 80
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.169, Regression, Logistic; Risk Difference (RD) = 0.14, 95% CI 2-sided [-0.06 to 0.35]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.001, Regression, Logistic; Risk Difference (RD) = 0.39, 95% CI 2-sided [0.15 to 0.63]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.002, Regression, Logistic; Risk Difference (RD) = 0.37, 95% CI 2-sided [0.14 to 0.60]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.59, 95% CI 2-sided [0.39 to 0.79]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.56, 95% CI 2-sided [0.34 to 0.78]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 0.57, 95% CI 2-sided [0.38 to 0.76]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p = 0.029, Regression, Logistic; Risk Difference (RD) = -0.23, 95% CI 2-sided [-0.44 to -0.02]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.898, Regression, Logistic; Risk Difference (RD) = 0.02, 95% CI 2-sided [-0.22 to 0.25]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.968, Regression, Logistic; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.24 to 0.23]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p = 0.033, Regression, Logistic; Risk Difference (RD) = 0.22, 95% CI 2-sided [0.02 to 0.42]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.099, Regression, Logistic; Risk Difference (RD) = 0.19, 95% CI 2-sided [-0.04 to 0.41]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p = 0.044, Regression, Logistic; Risk Difference (RD) = 0.20, 95% CI 2-sided [0.01 to 0.39]

6. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG)
Description: Change in FBG from baseline in LY3437943 relative to placebo and dulaglutide. LSMean was calculated using MMRM for post-baseline measures: Variable = Treatment*Time + Strata*Time + Baseline*Time.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
milligrams/deciliter (mg/dL) | -10.59 (5.98) | -46.26 (4.35) | -12.71 (6.95) | -30.19 (12.65) | -43.89 (8.42) | -66.09 (3.70) | -39.80 (10.79) | -65.20 (4.38)
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.823, Mixed Models Analysis; LSMean Difference = -2.12, 95% CI 2-sided [-20.73 to 16.48]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.165, Mixed Models Analysis; LSMean Difference = -19.60, 95% CI 2-sided [-47.29 to 8.10]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = -33.30, 95% CI 2-sided [-53.56 to -13.04]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -55.50, 95% CI 2-sided [-69.77 to -41.22]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.015, Mixed Models Analysis; LSMean Difference = -29.22, 95% CI 2-sided [-52.84 to -5.59]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -54.61, 95% CI 2-sided [-69.63 to -39.59]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 33.54, 95% CI 2-sided [18.26 to 48.82]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.231, Mixed Models Analysis; LSMean Difference = 16.07, 95% CI 2-sided [-10.25 to 42.39]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.804, Mixed Models Analysis; LSMean Difference = 2.37, 95% CI 2-sided [-16.28 to 21.01]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -19.83, 95% CI 2-sided [-31.01 to -8.65]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.586, Mixed Models Analysis; LSMean Difference = 6.45, 95% CI 2-sided [-16.75 to 29.65]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p = 0.002, Mixed Models Analysis; LSMean Difference = -18.94, 95% CI 2-sided [-30.93 to -6.96]

7. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG)
Description: Change in FBG from baseline in LY3437943 relative to placebo and dulaglutide. LSMean was calculated using MMRM for post-baseline measures: Variable = Treatment*Time + Baseline HbA1c Group (<=8.5%, >8.5%)*Time + Baseline BMI Group (<30kg/m2, >=30kg/m2)*Time + Baseline*Time.
Time Frame: Baseline, 36 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
mg/dL | -17.26 (10.87) | -27.53 (9.07) | -17.51 (5.59) | -21.46 (12.54) | -38.72 (10.81) | -69.10 (4.68) | -41.20 (14.43) | -67.84 (4.79)
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.984, Mixed Models Analysis; LSMean Difference = -0.25, 95% CI 2-sided [-24.57 to 24.07]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.804, Mixed Models Analysis; LSMean Difference = -4.20, 95% CI 2-sided [-37.44 to 29.03]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.167, Mixed Models Analysis; LSMean Difference = -21.47, 95% CI 2-sided [-51.91 to 8.98]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -51.84, 95% CI 2-sided [-76.09 to -27.59]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.168, Mixed Models Analysis; LSMean Difference = -23.94, 95% CI 2-sided [-57.94 to 10.06]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -50.58, 95% CI 2-sided [-74.94 to -26.22]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p = 0.362, Mixed Models Analysis; LSMean Difference = 10.02, 95% CI 2-sided [-11.55 to 31.60]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.696, Mixed Models Analysis; LSMean Difference = 6.07, 95% CI 2-sided [-24.34 to 36.48]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p = 0.436, Mixed Models Analysis; LSMean Difference = -11.19, 95% CI 2-sided [-39.38 to 16.99]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -41.57, 95% CI 2-sided [-62.89 to -20.25]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p = 0.418, Mixed Models Analysis; LSMean Difference = -13.67, 95% CI 2-sided [-46.75 to 19.42]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -40.31, 95% CI 2-sided [-60.77 to -19.85]

8. Secondary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline in LY3437943 relative to placebo and dulaglutide. LSMean was calculated using MMRM for post-baseline measures: Variable = Treatment*Time + Strata*Time + Baseline*Time.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
kilograms (kg) | -1.86 (0.66) | -1.16 (0.63) | -2.35 (0.48) | -6.27 (0.94) | -8.64 (1.23) | -11.99 (0.84) | -13.91 (1.38) | -12.84 (0.93)
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.540, Mixed Models Analysis; LSMean Difference = -0.49, 95% CI 2-sided [-2.07 to 1.08]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -4.41, 95% CI 2-sided [-6.69 to -2.13]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -6.78, 95% CI 2-sided [-9.47 to -4.09]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -10.13, 95% CI 2-sided [-12.24 to -8.03]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -12.06, 95% CI 2-sided [-15.06 to -9.06]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -10.99, 95% CI 2-sided [-13.24 to -8.73]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p = 0.135, Mixed Models Analysis; LSMean Difference = -1.19, 95% CI 2-sided [-2.75 to 0.37]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -5.11, 95% CI 2-sided [-7.36 to -2.86]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -7.48, 95% CI 2-sided [-10.19 to -4.77]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -10.83, 95% CI 2-sided [-12.89 to -8.77]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -12.76, 95% CI 2-sided [-15.74 to -9.77]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -11.69, 95% CI 2-sided [-13.90 to -9.47]

9. Secondary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline in LY3437943 relative to placebo and dulaglutide. LSMean was calculated using MMRM for post-baseline measures: Variable = Treatment*Time + Baseline HbA1c Group (<=8.5%, >8.5%)*Time + Baseline BMI Group (<30kg/m2, >=30kg/m2)*Time + Baseline*Time.
Time Frame: Baseline, 36 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 45 | 46 | 46 | 22 | 24 | 25 | 24 | 43
kilograms (kg) | -3.28 (0.92) | -1.97 (0.87) | -3.31 (0.62) | -7.28 (1.39) | -10.37 (1.49) | -16.48 (1.55) | -16.12 (1.63) | -17.18 (1.32)
Statistical Analysis 1: Comparison: Placebo vs 0.5 mg LY3437943; Test type: Superiority; p = 0.979, Mixed Models Analysis; LSMean Difference = -0.03, 95% CI 2-sided [-2.18 to 2.12]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.018, Mixed Models Analysis; LSMean Difference = -4.00, 95% CI 2-sided [-7.32 to -0.68]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -7.09, 95% CI 2-sided [-10.46 to -3.71]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -13.20, 95% CI 2-sided [-16.74 to -9.66]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -12.84, 95% CI 2-sided [-16.50 to -9.18]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -13.91, 95% CI 2-sided [-17.10 to -10.71]
Statistical Analysis 7: Comparison: 1.5 Milligram (mg) Dulaglutide vs 0.5 mg LY3437943; Test type: Superiority; p = 0.213, Mixed Models Analysis; LSMean Difference = -1.34, 95% CI 2-sided [-3.45 to 0.77]
Statistical Analysis 8: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (2 mg); Test type: Superiority; p = 0.002, Mixed Models Analysis; LSMean Difference = -5.31, 95% CI 2-sided [-8.66 to -1.97]
Statistical Analysis 9: Comparison: 1.5 Milligram (mg) Dulaglutide vs 4 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -8.40, 95% CI 2-sided [-11.76 to -5.04]
Statistical Analysis 10: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -14.51, 95% CI 2-sided [-18.00 to -11.01]
Statistical Analysis 11: Comparison: 1.5 Milligram (mg) Dulaglutide vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -14.15, 95% CI 2-sided [-17.77 to -10.54]
Statistical Analysis 12: Comparison: 1.5 Milligram (mg) Dulaglutide vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -15.22, 95% CI 2-sided [-18.36 to -12.07]

10. Secondary Outcome: Population PK: Average Steady-State Plasma Concentration (Cav,ss) of LY3437943
Description: The average steady-state plasma concentration of LY3437943 was evaluated using sparse sampling methodology/Population PK (PopPK) modeling.
Time Frame: Predose: Week 0, 1, 4, 12, 24, 30; Postdose: Week 2, 8, 16, 20, 36
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Number; unit: nanograms/milliliter (ng/mL)
Arm/Group | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 46 | 21 | 24 | 26 | 24 | 46
nanograms/milliliter (ng/mL) | 62.8 | 466 | 551 | 1100 | 1140 | 1620

ADVERSE EVENTS:
Time Frame: Baseline Through Study Completion (Up to 280 Days)
Description: All randomized participants who received at least one dose of study drug regardless of adherence to study drug or initiation of rescue medication. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 1.5 Milligram (mg) Dulaglutide | 0.5 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 (4 mg) | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46 | 0/47 | 0/23 | 0/24 | 0/26 | 0/24 | 0/46
Serious Adverse Events (participants affected / at risk) | 3/45 | 1/46 | 3/47 | 1/23 | 2/24 | 2/26 | 1/24 | 2/46
Other Adverse Events (participants affected / at risk) | 15/45 | 24/46 | 15/47 | 9/23 | 17/24 | 16/26 | 15/24 | 25/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=45) | 1.5 Milligram (mg) Dulaglutide (N=46) | 0.5 mg LY3437943 (N=47) | 4 mg LY3437943 (2 mg) (N=23) | 4 mg LY3437943 (4 mg) (N=24) | 8 mg LY3437943 (2 mg) (N=26) | 8 mg LY3437943 (4 mg) (N=24) | 12 mg LY3437943 (2 mg) (N=46)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1/22 (1) | 0/13 (0) | 0/24 (0) | 0/15 (0) | 0/12 (0) | 0/10 (0) | 0/9 (0) | 0/20 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=45) | 1.5 Milligram (mg) Dulaglutide (N=46) | 0.5 mg LY3437943 (N=47) | 4 mg LY3437943 (2 mg) (N=23) | 4 mg LY3437943 (4 mg) (N=24) | 8 mg LY3437943 (2 mg) (N=26) | 8 mg LY3437943 (4 mg) (N=24) | 12 mg LY3437943 (2 mg) (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3) | 2 (2) | 4 (5) | 3 (3) | 2 (2) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (2) | 2 (5) | 6 (7) | 5 (10) | 7 (9) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 3 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 8 (13) | 2 (2) | 2 (3) | 6 (9) | 7 (9) | 10 (15) | 9 (13)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 5 (11)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 3 (3)
Covid-19 (Infections and infestations) | 3 (3) | 4 (4) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (6)
Vaginal infection (Infections and infestations) | 0/23 (0) | 0/33 (0) | 0/23 (0) | 0/8 (0) | 0/12 (0) | 0/16 (0) | 1/15 (1) | 0/26 (0)
Lipase increased (Investigations) | 2 (2) | 1 (2) | 1 (1) | 1 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 2 (2) | 1 (1) | 5 (5) | 5 (5) | 4 (4) | 9 (9)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Penile swelling (Reproductive system and breast disorders) | 0/22 (0) | 1/13 (1) | 0/24 (0) | 0/15 (0) | 0/12 (0) | 0/10 (0) | 0/9 (0) | 0/20 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/23 (0) | 0/33 (0) | 0/23 (0) | 0/8 (0) | 0/12 (0) | 1/16 (2) | 0/15 (0) | 0/26 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT04867785/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT04867785/SAP_001.pdf